CLINICAL TRIAL: NCT00378521
Title: Phase II Dose Response Study of a Topical Gel Formulation of Nitroglycerin, MQX-503, in the Treatment of Raynaud's Phenomenon
Brief Title: Dose Response Study of a Topical Gel for the Treatment of Raynaud's Phenomenon
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MediQuest Therapeutics (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 06-001
Record Dates: First submitted 2006-09-18; First posted 2006-09-20 (Estimated); Last update posted 2007-05-30 (Estimated); Status verified 2007-05

CONDITIONS: Raynaud's Disease; Raynaud's Disease Secondary to Scleroderma; Raynaud's Disease Secondary to Autoimmune Disease
Keywords: Raynaud's; Nitroglycerin; topical gel; cold hands; painful hands; scleroderma
MeSH Terms: conditions — Raynaud Disease; Scleroderma, Diffuse

INTERVENTIONS:
Drug: MQX-503

SUMMARY:
The Purpose of this study is to determine the response to two different strengths of a topical gel containing nitroglycerin in patients with Raynaud's disease.

DETAILED DESCRIPTION:
The Purpose of this clinical study is to determine, in a controlled fashion, the response to two dosage strengths of a topical gel formulation of Nitroglycerin, MQX-503, in the determination of changes in finger blood flow and skin temperature in the fingers of patients with moderate to severe primary Raynaud's phenomenon and with Raynaud's phenomenon secondary to autoimmune diseases, such as scleroderma. The dosage strength response in the treatment of the symptoms (pain, tingling, numbness) will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients, 18 to 75 years
* Clinical Diagnosis of Raynaud's, or observed event by study physician, or symptoms with reduced blood flow as meausred using laser doppler equipment
* Agree to have test gels applied to finger
* Discontinue current vasodialator therapeis for Raynaud's treatment
* Four weeks from last clinical trial participation
* Agree not to use any other investigational medications or therapies to treat Raynaud's and its symptoms while participating in this study including other dosages or forms of nitroglycerin, isosorbide dinitrate, fenoldopam mesylate, milrinone lactate, nifedipine, diltiazem, felodipine, nimodipine, nisoldipine, and verapamil
* Negative pregnancy test for women prior to study start and agree to use effective contraception throughout
* Must be able to give written informed consent and comply with all study requirements

Exclusion Criteria:

* Concurrent use of any nitrate medication or medications known to interact with Nitroglycerin such as sildenafil, and other treatments for erectile dysfunction
* Patients who have a known allergy to Nitroglycerin or common topical gel ingredients
* Patients with a history of migraine, cluster or vascular headaches, or those who suffer from chronic pain
* Patients with a history of an unstable medical problem or any current condition that would interfere in participation in the study
* Patients unable to complete pain assessment instructions
* Patients who in the last three months have had a myocardial infarction, uncontrolled congestive heart failure, unstable angina, uncontrolled hypotension or uncontrolled hypertension
* Patients who have participated in another investigational drug study within four weeks of the first study treatment
* Patients with out of range laboratory screening values
* Patients who have had major abdominal, thoracic or vascular surgery within six months of the first study treatment
* Patients with open lesions or skin conditions where gel is to be applied
* Pregnant or nursing women
* Women who will not agree to comply with contraceptive requirements
* Patients with a history of poor compliance, poor cooperation or unreliability

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2006-07; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Measure the time required for blood flow to return to baseline after cold exposure

SECONDARY OUTCOMES:
Measure the time required for skin temperature to return to baseline after cold exposure
Prevention or reduction of symptoms following cold exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Klaff, MD, Principal Investigator — Rainier Clinical Research
Locations (1):
- Rainier Clinical Research, Renton, Washington, United States